CLINICAL TRIAL: NCT02129764
Title: Prednisone in Uric Acid Lowering in Symptomatic Heart Failure PATients With Hyperuricemia (PUSH-PATH Study 2)
Brief Title: Prednisone for Heart Failure Patients With Hyperuricemia
Acronym: PUSH-PATH-2
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Hebei Medical University (Other)
Responsible Party: Principal Investigator, Kun-shen Liu M.D., Professor, Hebei Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUSH-PATH 2
Record Dates: First submitted 2014-04-30; First posted 2014-05-02 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Heart Failure, Hyperuricemia
MeSH Terms: conditions — Heart Failure; Hyperuricemia | interventions — Prednisone; Allopurinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prednisone (Experimental): Prednisone will be given 30mg/day for 2 weeks and then tapered off.
  Interventions: Drug: Prednisone
- Allopurinol (Active Comparator): Allopurinol will be given 100 mg/day initially, and then titrated to 200 mg/day.
  Interventions: Drug: Allopurinol

INTERVENTIONS:
Drug: Prednisone
  Arms: Prednisone
Drug: Allopurinol
  Arms: Allopurinol

SUMMARY:
Hyperuricemia is a very common finding in patients with heart failure. It is usually related to diuretic use and deteriorated renal function. The recently evidence showed that prednisone and allopurinol may have similar effect on uric acid (UA) lowering in symptomatic heart failure patients with hyperuricemia, but prednisone may be superior over allopurinol in renal function improvement. Thus the investigators design this randomized head to head study to test their hypothesis that prednisone is superior over allopurinol in renal function improvement despite their similar effect on UA lowering in heart failure patients with hyperuricemia.

DETAILED DESCRIPTION:
Hyperuricemia in heart failure (HF) is linked to renal impairment, hemodynamic compromise, and inflammation. Hyperuricemic HF patients are characterized by worsening of renal function and fragile volume state, both of which restrict the use of non-steroidal anti-inflammatory drugs (NSAIDs) when treating concurrent inflammatory diseases. Recent small studies suggest that steroidal anti-inflammatory drug, prednisone, may have renal protective, UA lowering, and potentiating diuretic effects in hyperuricemic HF patients. However, general acceptance of prednisone as a treatment option for anti-inflammation therapy in patients with hyperuricemic HF requires more safety data. We therefore designed a randomized study to compare the safety and renal protective effects of short-term use of prednisone with allopurinol, a widely used xanthine oxidase inhibitor with a well-established safety profile in HF, in hyperuricemic HF patients.

ELIGIBILITY:
Inclusion Criteria:

* chronic congestive heart failure
* 18-80 years old
* NYHA Class II-IV
* Serum uric acid > 7mg/dl
* left ventricular ejection fraction ≤ 45%

Exclusion Criteria:

* Acute gouty arthritis;
* Any condition (other than heart failure) that could limit the use of prednisone or xanthine oxidase inhibitors;
* Acute decompensated heart failure;
* Any concurrent disease that likely limits life expectancy;
* Active myocarditis, or an hypertrophic obstructive or restrictive cardiomyopathy;
* Myocardial infarction, stroke, unstable angina, or cardiac surgery within the previous 3 months;
* Indication for hemodialysis
* Creatinine> 3.0 mg per deciliter at admission to the hospital
* Uncontrolled systolic blood pressure > 140 mmHg
* Known bilateral renal artery stenosis
* Complex congenital heart disease
* Any signs of infections
* Enrollment in another clinical trial involving medical or device-based interventions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in serum creatinine levels | 2 weeks
  Change from baseline in serum creatinine levels at the end of study, i.e. 2 weeks

SECONDARY OUTCOMES:
Change from baseline in uric acid levels | 2 weeks
  Change from baseline in uric acid levels at the end of study, i.e. 2 weeks
Change from baseline in Cystatin C | 2 weeks
  Change from baseline in cystatin c at the end of study, i.e. 2 weeks.
the levels of tumor necrosis factor (TNF) alfa,IL-6 in the circulation, high-sensitivity C-reactive Protein (hs-CRP) | 2 weeks
  Change of plasma TNF-alfa, IL-6, and hs-CRP levels at the end of study, i.e. 2 weeks (expressed as percentage of baseline)
The levels of angiotensin II and aldosterone in the circulation. | 2 weeks
  Change of plasma angiotensin II and aldosterone at end of week-1 (i.e. on day 7) and at the end of week-2 (i.e. on day 14), the values were expressed as percentage of baseline)
Daily urine output | 2 weeks
  24-hour urine output at week-1 (i.e. on day 7) and at week-2 (i.e. on day 14)
New York Heart Association (NYHA) functional class | 2 weeks
  Change of NHHA functional class at the end of study
24h urinary sodium excretion | 2 weeks
  24-hour urinary sodium excretion at week-1 (i.e. on day 7) and at week-2 (i.e. on day 14)

CONTACTS AND LOCATIONS:
Locations (1):
- Shijiazhuang, Hebei, China